CLINICAL TRIAL: NCT01111409
Title: A Prospective, Multi-Centre Pilot Study to Evaluate the Clinical Effectiveness and Safety of the VFIX Device as Treatment for Apical Prolapse
Brief Title: A Pilot Study to Evaluate the Clinical Effectiveness and Safety of the VFIX Device as Treatment for Apical Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 300-08-013
Record Dates: First submitted 2010-04-26; First posted 2010-04-27 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2011-12

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VFIX (Experimental)
  Interventions: Device: VFIX Device

INTERVENTIONS:
Device: VFIX Device — Sterile, single-use instrument capable of delivering an absorbable PDS suture anchor

SUMMARY:
The primary objective of this pilot study is to evaluate the safety and effectiveness of the VFIX device in maintaining vaginal apical support for at least 6 months in women with symptomatic apical prolapse (upper vaginal or uterine prolapse).

DETAILED DESCRIPTION:
Assuming success of the VFIX anatomical observational study (protocol 300-08-009), in this pilot study approximately 20 subjects (excluding the Device Run-In (DRI) subjects) will undergo the VFIX procedure to evaluate the safety and effectiveness of the VFIX device in maintaining apical support for at least 6 months, in women with symptomatic apical prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Subjects of child bearing potential have a negative blood or urine pregnancy test prior to the procedure and subject has completed childbearing
* Subject with apical prolapse at stage II or more and requiring treatment (C should be at least -1 cm)
* On reduction of the apical prolapse, leading edge of prolapse should be at or above the hymen
* If applicable, subject has small/normal size uterus and there is no elongation of the cervix as determined by clinical assessment
* The vaginal apex can reach the Sacrospinous Ligament (SSL) on exam
* Subjects are allowed concurrent incontinence procedure as required
* Concurrent perineal repairs and excision of excess vaginal tissue repairs as required
* Agrees to participate in the study, including completion of all study-related procedures, evaluations and questionnaires, and documents this agreement by signing the Ethics Committee approved informed consent

Exclusion Criteria:

* Additional surgical intervention for POP repairs concurrent to the VFIX procedure (including, but not limited to sacrocolpopexy, paravaginal repair, colporrhaphy, mesh repair, etc)
* Experimental drug or experimental medical device within 3 months prior to the planned procedure
* Active genital, urinary or systemic infection at the time of the surgical procedure. Surgery may be delayed in such subjects until the infection is cleared.
* Previous hysterectomy within 6 months of scheduled surgery.
* Coagulation disorder or on therapeutic anticoagulant therapy (except aspirin) at the time of surgery
* Nursing or pregnant
* Presence of cancers of the vagina, cervix, or uterus
* In the investigator's opinion, any medical condition or psychiatric illness that could potentially be life threatening or affect their ability to complete the study visits according to this protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2010-11 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Robinson, MD, Study Director — Ethicon, Inc.
Locations (3):
- Australia (3):
  - QEII Hospital, Brisbane
  - Frances Perry House, Parkville
  - Urogynaecology Unit, Royal Women's Hospital, Parkville